CLINICAL TRIAL: NCT03661762
Title: Production of a Device to Obtain Continuous Ambulatory Vestibular Assessment (CAVA) - Healthy Volunteer Trial
Acronym: CAVA
Status: Completed | Type: Observational
Sponsor: Julie Dawson (Other)
Collaborators: University of East Anglia (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor-Investigator, Julie Dawson, Manager Research Services, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Other Study IDs: 240847 (28-02-18)
Record Dates: First submitted 2018-07-26; First posted 2018-09-07 (Actual); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Optokinetic Nystagmus
Keywords: eye movements; electronystagmography; nystagmus; electrooculogram; vestibular assessment
MeSH Terms: conditions — Nystagmus, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: All trial participants are within this group. All trial participants will wear the CAVA device for up to 23 hours a day, for 30 days.
  Interventions: Device: CAVA

INTERVENTIONS:
Device: CAVA — prototype device for monitoring dizziness

SUMMARY:
Clinical investigation of a medical device (CAVA) for recording eye movements. Healthy volunteers will wear the device for 23 hours a day, for 30 days. On 8 separate days of the trial they will induce optokinetic nystagmus (a normal reflex in response to full-field motion) by watching a short video of less than 1 minute in duration. The data will be analysed offline by a scientist, who will attempt to identify the dates that the nystagmus was induced.

DETAILED DESCRIPTION:
Dizziness is a common condition that is responsible for a significant degree of material morbidity and burden on the National Health Service. There are multiple causes of dizziness, and these originate from pathologies affecting a large variety of different organ systems. Dizziness is usually episodic and short-lived, so when a patient presents to their health care provider, examination is often normal. As such, diagnosis is challenging and patients often experience significant delay in receiving a diagnosis. The investigators have developed a prototype device for monitoring dizziness and have tested it in a small group of volunteers. The results showed that their device is capable of accurately, precisely and reliably identifying periods of dizziness over a short period of time. Independent market research has confirmed that their device could meet the required clinical need, would be desired by clinicians, and that there is no equivalent solution currently available. The investigators have received an award from the Medical Research Council to trial their device in a large cohort of healthy volunteers. Once completed, they will be positioned well to test their device in a cohort of patients with a defined dizziness syndrome, before further testing their device in a more diverse patient population. Once validated, developed and brought to market, the device would provide early diagnosis and accurate treatment for a significant proportion of the patient population. This would save the National Health Service money by reducing multiple visits to General Practitioner clinics, reducing referrals to multiple specialist clinics, and reducing treatment required from falls and other conditions associated with dizziness.

The overall aim of this trial is to test a fully evolved device for the continuous recording of eye movements over a prolonged period of time. For the purpose of this study, the monitoring period is 23 hours a day, for 30 days. The device is composed of two components: a bespoke single-use sensor array that adheres to the participant's face, and a small reusable module that contains a battery, microcomputer, data storage facility, battery and connection port.

The investigators intend to confirm that the device will be able to capture any occurrence, of a minimum period of thirty seconds, of artificially induced nystagmus, within a 24-hour period of time. Each participant will be provided with the device and enough single-use electrode arrays to allow the array to be changed every 24 hours, for thirty days. Participants will be allowed to remove the sensor array for up to 60 minutes each day to allow them to wash and/or shower. On eight of the thirty days for which they wear the array, each participant will be required to induce physiological nystagmus by viewing optokinetic video footage. The footage will be viewed on a portable screen (of a deactivated mobile phone) inside a Virtual Reality headset. These will be issued to the participants at the beginning of the trial. Participants will undertake the procedure whilst stationary for the first four days, and whilst walking gently on the spot for the remaining four days. The identity of these days will not be revealed to the blinded investigator who will later analyse the data. At the end of the thirty-day trial, the sensitivity and specificity of the device will be determined by assessing whether the data can be used to correctly identify the dates that participants induced nystagmus.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over
* Able to commit to 30 days of continuous wear of the trial device as per the study plan
* Own a telephone

Exclusion Criteria:

* Potential participants who have a history of dermatological disease or damage around the forehead
* Potential participants who have an allergy to plasters and/or medical adhesives
* History of dizziness, vertigo, balance disorders, or syncope
* History of hypertension or cardiac problems (uncontrolled, acute or de-compensated phase)
* History of ear disease, or previous ear surgery
* History of psychotic/neurotic disorders or epilepsy
* History of eye disease, or previous eye surgery
* Unable to follow the testing protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, aged 18 or over.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Phillips, Consultant, Principal Investigator — Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK)
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 18
Completed | 10
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Healthy Volunteers [Count of Participants; unit: Participants] — All genders over 18 years of age.
  Participants | 18

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of a Computer Algorithm to Detect Artificially Induced Nystagmus
Description: Dates containing nystagmus. Of the ~450 days' worth of data captured during the study, 120 will contain artificially induced nystagmus. A computer algorithm has been developed at the University of East Anglia for detecting nystagmus. The key measurements are the sensitivity and specificity of the algorithm's results when applied to data captured during the trial. This measurement will be assessed post-trial.
Time Frame: 30 days
Measure: Number; unit: Percent
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 17
Percent
  Sensitivity | 99.1
  Specificity | 98.6

2. Secondary Outcome: Post-trial Participant Questionnaire.
Description: A 2-page questionnaire producing qualitative and quantitative data. Participants rate different aspects of their experiences with the device using a sliding scale and have the opportunity to write more detailed descriptions.
Time Frame: 30 days
Reporting Status: Not Posted

3. Secondary Outcome: Compliance With the Device.
Description: 1 - There is a minimum of 80% compliance with wearing the device for each single day of the trial for a minimum of 80% of participants. 2 There is a minimum of 80% compliance with wearing the device for the entirety of the 30-day trial for a minimum of 80% of participants.
Time Frame: 30 days
Population: For the 30-day trial compliance, the number of participants differs as not all participants completed the trial in full.
Measure: Number; unit: percentage of participants
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 17
percentage of participants
  Daily compliance | 82
  30-day compliance: number analyzed (Participants) | 10
  30-day compliance | 100

4. Secondary Outcome: Data Usefulness
Description: The device provides less than 5% non-useful data for each participant. We will report the percentage of non-useful data (corrupted or flat-line data) that is captured for each participant.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Percentage of non-useful data
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 17
Percentage of non-useful data | 0 (0)

5. Secondary Outcome: Data Usefulness
Description: The device provides less than 5% non-useful data for the entirety of the 30-day trial across all participants. We will report the percentage of non-useful data (corrupted or flat-line data) that is captured over the entire trial, across all participants.
Time Frame: 30 days
Measure: Number; unit: percentage of non-useful data
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 17
percentage of non-useful data | 0

6. Secondary Outcome: Event Marker Functioning
Description: During a return visit, the event marker on each device will be pressed and the time noted. Post-trial, the data on the device will be examined to confirm that an event was recorded on the correct date. This will produce either a positive or negative outcome, depending on whether the event marker button press is present in the data or not. The percentage of identifiable button presses across all devices will be reported.
Time Frame: 30 days
Measure: Number; unit: percentage of button presses identified
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 17
percentage of button presses identified | 100

7. Secondary Outcome: Time Stamp Accuracy
Description: The difference will be calculated between the time noted by the research team and the time logged by the device when the event marker was activated. The time difference (in hh:mm:ss) will be calculated across all devices and we will report the average and standard deviation of the clock drift.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 17
minutes per day | -17.49 (1.47)

8. Secondary Outcome: Accelerometer Functioning
Description: Participants will perform a number of head movements and the device data will be examined visually to confirm that they can be identified. This will produce either a positive or negative outcome for each head movement, depending on whether the movement is visible in the data or not. The proportion of successfully identified head movements will be reported.
Time Frame: 30 days
Measure: Number; unit: percentage of movements identified
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 17
percentage of movements identified
  Slow head turning | 97
  Slow head nodding | 100
  Slow head tilting | 100
  Fast head turning | 93
  Fast head nodding | 100
  Fast head tilting | 97

9. Secondary Outcome: Accuracy of Nystagmus Beat Direction
Description: Participants will undergo caloric testing at the end of the trial, during which they will wear conventional Videonystagmography (VNG) goggles as well as the CAVA device. The beat direction (whether the fast phase of the nystagmus is towards the left or right ear) will be determined from both sources of data during the period of nystagmus captured. This will produce either a positive or negative outcome, depending on whether the beat direction matches in both data sources. The proportion of matches will be reported.
Time Frame: 1 hour
Reporting Status: Not Posted

10. Secondary Outcome: Accuracy of Nystagmus Onset Time
Description: Also from the data captured during caloric testing, the start time of nystagmus will be identified from both the VNG data and data captured by the CAVA device. The time difference (in mm:ss) will be calculated between the two data sources and the mean time difference will be reported.
Time Frame: 1 hour
Reporting Status: Not Posted

11. Secondary Outcome: Accuracy of Nystagmus Finishing Time
Description: Also from the data captured during caloric testing, the finishing time of nystagmus will be identified from both the VNG data and data captured by the CAVA device. The time difference (in mm:ss) will be calculated between the two data sources and the mean time difference will be reported.
Time Frame: 1 hour
Reporting Status: Not Posted

12. Secondary Outcome: Accuracy of Nystagmus Peak Time
Description: Also from the data captured during caloric testing, the time at which the nystagmus reaches its maximum slow phase velocity will be calculated from the VNG data and the data captured by the CAVA device. The time difference (in mm:ss) will be calculated between the two data sources and the mean time difference will be reported.
Time Frame: 1 hour
Reporting Status: Not Posted

13. Secondary Outcome: Accuracy of Nystagmus Frequency
Description: Also from the data captured during caloric testing, the number of beats will be counted during the period identified as the nystagmus peak time. This will be calculated for both the VNG data and the data captured by the CAVA device. From the number of beats and time duration examined, the frequency of the nystagmus will be determined. The difference between the two systems will be calculated and the mean difference will be reported. The Unit of Measure will be Hz (number of beats per second).
Time Frame: 1 hour
Reporting Status: Not Posted

14. Secondary Outcome: Data Drop-outs
Description: The device provides less 5 drop-outs for each single day of the trial for each participant. We will report the maximum number of drop-outs (periods when the device stopped logging) per participant, per day.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Number of drop outs
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 17
Number of drop outs | 0.2353 (0.4372)

15. Secondary Outcome: Data Drop-outs
Description: The device provides less 60 drop-outs for the entirety of the 30-day trial across all participants. We will report the total number of drop-outs that occurred over the entire trial, across all participants.
Time Frame: 30 days
Population: Healthy volunteers
Measure: Number; unit: Total number of drop outs
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 17
Total number of drop outs | 4

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 10/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers (N=18)
Over rubbed under left eye (Skin and subcutaneous tissue disorders) | 1 (1)
Erosion under all electrode sites (Skin and subcutaneous tissue disorders) | 1 (1)
Redness under electrodes (Skin and subcutaneous tissue disorders) | 8 (8)
Disturbed sleep (Product Issues) | 1 (1) — Participant had difficulty sleeping whilst wearing the device for several days
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) — This adverse event was deemed to be unrelated to the study
Allergic reaction (Skin and subcutaneous tissue disorders) | 1 (1) — Participant experienced an allergic reaction to the materials used in the device's electrode pads
Swollen lymph nodes (Respiratory, thoracic and mediastinal disorders) | 1 (1) — This adverse event was deemed to be unrelated to the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT03661762/Prot_SAP_000.pdf